CLINICAL TRIAL: NCT01545232
Title: Pragmatic, Randomized Optimal Platelet and Plasma Ratios
Acronym: PROPPR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Resuscitation Outcomes Consortium (Network); Defence Research and Development Canada (Industry)
Responsible Party: Principal Investigator, John Holcomb, Study Director, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-GEN-11-0174; U01HL077863 (NIH)
Record Dates: First submitted 2012-02-29; First posted 2012-03-06 (Estimated); Results first posted 2015-06-03 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Trauma
Keywords: Massive Transfusion; Trauma; Coagulopathy; Trauma Induced Coagulopathy; Plasma; Platelets; Red Blood Cells; Mortality; Wounds and Injuries; Shock, Hemorrhagic; Shock; Pathologic Processes; Hemorrhage; Hemostatics; Coagulation; Transfusion-related acute lung injury (TRALI); Inflammation
MeSH Terms: conditions — Wounds and Injuries; Hemostatic Disorders; Shock, Hemorrhagic; Shock; Pathologic Processes; Hemorrhage; Thrombosis; Transfusion-Related Acute Lung Injury; Inflammation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1:1:1 Blood Transfusion Ratio (Active Comparator)
  Interventions: Biological: 1:1:1 Blood Transfusion Ratio
- 1:1:2 Blood Transfusion Ratio (Active Comparator)
  Interventions: Biological: 1:1:2 Blood Transfusion Ratio

INTERVENTIONS:
Biological: 1:1:1 Blood Transfusion Ratio — Group 1 will be randomized to receive the 1:1:1 ratio of plasma:platelets:RBC. Blood bank will prepare the initial container containing 6 units plasma, 1 unit platelets (a pool of 6 units on average) and 6 units RBC; the blood bank will send the initial and all subsequent containers until notified of the discontinuation of the PROPPR transfusion protocol.
  Arms: 1:1:1 Blood Transfusion Ratio
Biological: 1:1:2 Blood Transfusion Ratio — Group 2 will be randomized to receive the 1:1:2 ratio of plasma:platelets:RBC. The blood bank will prepare the initial container containing 3 units plasma, 0 units platelets and 6 units RBC, a second container containing 3 units plasma, 1 unit platelets (a pool of 6 units on average) and 6 units RBC, and the blood bank will send this sequence of 2 containers repeatedly, until notified of the discontinuation of the PROPPR transfusion protocol.
  Arms: 1:1:2 Blood Transfusion Ratio

SUMMARY:
Pragmatic, Randomized, Optimal Platelet and Plasma Ratios (PROPPR)is a Phase III trial designed to evaluate the difference in 24-hour and 30-day mortality among subjects predicted to receive massive transfusion ([MT] (defined as receiving 10 units or more red blood cells (RBCs) within the first 24 hours). The goal of PROPPR is to improve the basis on which clinicians make decisions about transfusion protocols for massively bleeding patients.

PROPPR is a Resuscitation Outcomes Consortium (ROC) Protocol. ROC is funded by the National Heart, Lung, and Blood Institute (NHLBI), the United States' Department of Defense (DoD) and the Defence Research and Development Canada. PROPPR will be conducted as a Phase III trial at Level I Adult Trauma Centers in North America.

DETAILED DESCRIPTION:
Background: Multiple observational studies have reported that blood product component ratios (i.e., plasma:platelets:RBCs) that approach the 1:1:1 ratio, found in fresh whole blood, are associated with significant decreases in truncal hemorrhagic death and in overall 24-hour and 30-day mortality among injured patients. The rationale for the 1:1:1 ratio is that the closer a transfusion regimen approximates whole blood, the faster hemostasis will be achieved with minimum risk of coagulopathy. The current DoD guideline specifies the use of 1:1:1, and this practice is followed on almost all combat casualties. In other observational studies, leading centers have reported good outcomes across a range of different blood product ratios. For example, a 1:2 plasma:RBC ratio is used with little guidance regarding platelets. The proposed randomized trial is intended to resolve debate and uncertainty regarding optimum blood product ratios.

Study Design: Randomized, two-group, controlled Phase III trial with a Vanguard stage. Equal random allocation to treatment using stratified, permuted blocks with randomly chosen block sizes and stratification by site.

Objective: To conduct a Phase III multi-site, randomized trial in subjects predicted to have a massive transfusion, comparing the efficacy and safety of 1:1:1 transfusion ratios of plasma and platelets to red blood cells (the closest approximation to reconstituted whole blood) with the 1:1:2 ratio. The co-primary outcomes will be 24-hour and 30-day mortality. The PROPPR Trial will be conducted with exception from informed consent (EFIC). Additionally, laboratory data from the trial will add to the understanding of trauma induced coagulopathy (TIC) and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who require the highest trauma team activation at each participating center,
* Estimated age of 15 years or older or greater than/equal to weight of 50 kg if age unknown,
* Received directly from the injury scene,
* Initiated transfusion of at least one unit of blood component within the first hour of arrival or during prehospital transport, and
* Predicted to receive a MT by exceeding the threshold score of either the Assessment of Blood Consumption (ABC) score or the attending trauma physician's judgment criteria

Exclusion Criteria:

* Received care (as defined as receiving a life saving intervention) from an outside hospital or healthcare facility (Procedures and care given at an outside health facility cannot be documented or controlled resulting in a high variability of standards of care and clinical outcomes.)
* Moribund patient with devastating injuries and expected to die within one hour of Emergency Department (ED) admission
* Prisoners, defined as those who have been directly admitted from a correctional facility
* Patients requiring an emergency thoracotomy
* Children under the age of 15 years or under 50 kg body weight if age unknown
* Known pregnancy in the ED
* Greater than 20% total body surface area (TBSA) burns
* Suspected inhalation injury
* Received greater than five consecutive minutes of cardiopulmonary resuscitation (CPR with chest compressions) in the pre-arrival or ED setting
* Known Do Not Resuscitate (DNR) prior to randomization
* Enrolled in a concurrent, ongoing interventional, randomized clinical trial
* Patients who have activated the "opt-out" process or patients/legally authorized representatives that refuse blood products on arrival to ED.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 680 (Actual)
Dates: Start 2012-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Holcomb, MD, Study Director — The University of Texas Health Science Center, Houston
Locations (12):
- United States (11):
  - University of Alabama, Birmingham, Alabama
  - University of Arizona, Tucson, Arizona
  - University of Southern California, Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - University of Maryland School of Medicine, Baltimore, Maryland
  - University of Cincinnati, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - University of Texas Health Science Center- Memorial Hermann Hospital, Houston, Texas
  - University of Washington- Harborview Medical Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Sunnybrook Health Science Center, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Levy DT, Livingston CE, Saroukhani S, Fox EE, Wade CE, Holcomb JB, Gumbert SD, Galvagno SM Jr, Kaslow OY, Pittet JF, Pivalizza EG. Association of Opioid Administration During General Anesthesia and Survival for Severely Injured Trauma Patients: A Preplanned Secondary Analysis of the PROPPR Study. Anesth Analg. 2023 May 1;136(5):905-912. doi: 10.1213/ANE.0000000000006456. Epub 2023 Apr 14. PMID 37058726
- [Derived] McCully BH, Wade CE, Fox EE, Inaba K, Cohen MJ, Holcomb JB, Schreiber MA; PROPPR study group. Temporal profile of the pro- and anti-inflammatory responses to severe hemorrhage in patients with venous thromboembolism: Findings from the PROPPR trial. J Trauma Acute Care Surg. 2021 May 1;90(5):845-852. doi: 10.1097/TA.0000000000003088. PMID 33797501
- [Derived] DeSantis SM, Brown DW, Jones AR, Yamal JM, Pittet JF, Patel RP, Wade CE, Holcomb JB, Wang H; PROPPR Study Group. Characterizing red blood cell age exposure in massive transfusion therapy: the scalar age of blood index (SBI). Transfusion. 2019 Aug;59(8):2699-2708. doi: 10.1111/trf.15334. Epub 2019 May 3. PMID 31050809
- [Derived] Jones AR, Patel RP, Marques MB, Donnelly JP, Griffin RL, Pittet JF, Kerby JD, Stephens SW, DeSantis SM, Hess JR, Wang HE; PROPPR Study Group. Older Blood Is Associated With Increased Mortality and Adverse Events in Massively Transfused Trauma Patients: Secondary Analysis of the PROPPR Trial. Ann Emerg Med. 2019 Jun;73(6):650-661. doi: 10.1016/j.annemergmed.2018.09.033. Epub 2018 Nov 15. PMID 30447946
- [Derived] Cardenas JC, Zhang X, Fox EE, Cotton BA, Hess JR, Schreiber MA, Wade CE, Holcomb JB; PROPPR Study Group. Platelet transfusions improve hemostasis and survival in a substudy of the prospective, randomized PROPPR trial. Blood Adv. 2018 Jul 24;2(14):1696-1704. doi: 10.1182/bloodadvances.2018017699. PMID 30030268
- [Derived] Henry B, Perez A, Trpcic S, Rizoli S, Nascimento B. Protecting study participants in emergency research: is community consultation before trial commencement enough? Trauma Surg Acute Care Open. 2017 Jul 12;2(1):e000084. doi: 10.1136/tsaco-2017-000084. eCollection 2017. PMID 29766088
- [Derived] Galvagno SM Jr, Fox EE, Appana SN, Baraniuk S, Bosarge PL, Bulger EM, Callcut RA, Cotton BA, Goodman M, Inaba K, O'Keeffe T, Schreiber MA, Wade CE, Scalea TM, Holcomb JB, Stein DM; PROPPR Study Group. Outcomes after concomitant traumatic brain injury and hemorrhagic shock: A secondary analysis from the Pragmatic, Randomized Optimal Platelets and Plasma Ratios trial. J Trauma Acute Care Surg. 2017 Oct;83(4):668-674. doi: 10.1097/TA.0000000000001584. Epub 2017 Jun 6. PMID 28930959
- [Derived] Naumann DN, Vincent LE, Pearson N, Beaven A, Smith IM, Smith K, Toman E, Dorrance HR, Porter K, Wade CE, Cotton BA, Holcomb JB, Midwinter MJ. An adapted Clavien-Dindo scoring system in trauma as a clinically meaningful nonmortality endpoint. J Trauma Acute Care Surg. 2017 Aug;83(2):241-248. doi: 10.1097/TA.0000000000001517. PMID 28731937
- [Derived] Holcomb JB, Tilley BC, Baraniuk S, Fox EE, Wade CE, Podbielski JM, del Junco DJ, Brasel KJ, Bulger EM, Callcut RA, Cohen MJ, Cotton BA, Fabian TC, Inaba K, Kerby JD, Muskat P, O'Keeffe T, Rizoli S, Robinson BR, Scalea TM, Schreiber MA, Stein DM, Weinberg JA, Callum JL, Hess JR, Matijevic N, Miller CN, Pittet JF, Hoyt DB, Pearson GD, Leroux B, van Belle G; PROPPR Study Group. Transfusion of plasma, platelets, and red blood cells in a 1:1:1 vs a 1:1:2 ratio and mortality in patients with severe trauma: the PROPPR randomized clinical trial. JAMA. 2015 Feb 3;313(5):471-82. doi: 10.1001/jama.2015.12. PMID 25647203
- [Derived] Baraniuk S, Tilley BC, del Junco DJ, Fox EE, van Belle G, Wade CE, Podbielski JM, Beeler AM, Hess JR, Bulger EM, Schreiber MA, Inaba K, Fabian TC, Kerby JD, Cohen MJ, Miller CN, Rizoli S, Scalea TM, O'Keeffe T, Brasel KJ, Cotton BA, Muskat P, Holcomb JB; PROPPR Study Group. Pragmatic Randomized Optimal Platelet and Plasma Ratios (PROPPR) Trial: design, rationale and implementation. Injury. 2014 Sep;45(9):1287-95. doi: 10.1016/j.injury.2014.06.001. Epub 2014 Jun 10. PMID 24996573
- [Derived] Lissauer ME, Galvagno SM Jr, Rock P, Narayan M, Shah P, Spencer H, Hong C, Diaz JJ. Increased ICU resource needs for an academic emergency general surgery service*. Crit Care Med. 2014 Apr;42(4):910-7. doi: 10.1097/CCM.0000000000000099. PMID 24335442

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1:1:1 Blood Transfusion Ratio | 1:1:2 Blood Transfusion Ratio
Started | 338 | 342
Completed | 338 | 342
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1:1:1 Blood Transfusion Ratio | 1:1:2 Blood Transfusion Ratio | Total
Number analyzed (Participants) | 338 | 342 | 680
Age, Customized [Number; unit: participants] — 15 years of age or older
  participants | 338 | 342 | 680
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 59 | 134
  Male | 263 | 283 | 546
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 61 | 59 | 120
  Not Hispanic or Latino | 277 | 283 | 560
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 2 | 8
  Asian | 21 | 8 | 29
  Native Hawaiian or Other Pacific Islander | 3 | 1 | 4
  Black or African American | 93 | 93 | 186
  White | 210 | 224 | 434
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 3 | 14 | 17

OUTCOME MEASURES:

1. Primary Outcome: 24-hour Mortality
Time Frame: First 24 hours after ED admission
Population: Number of subjects who were randomized to each group
Measure: Number; unit: participants
Arm/Group | 1:1:1 Blood Transfusion Ratio | 1:1:2 Blood Transfusion Ratio
Number analyzed (Participants) | 338 | 342
participants | 43 | 58
Statistical Analysis 1: Comparison: 1:1:1 Blood Transfusion Ratio vs 1:1:2 Blood Transfusion Ratio; Initial sample size (580) planned to detect a clinically meaningful 10% difference in 24-hour mortality (11% vs. 21%) supported by prior data. Data Safety Monitoring Board (DSMB) increased sample size to 680 according to trial's adaptive design. With 680 pts. & given the final observed mortality proportions in 1:1:1 group, PROPPR had 95% power to detect the pre-specified 10% difference at 24 hours if such differences existed; Test type: Superiority or Other; p = 0.12, Mantel Haenszel; The critical level for significance (p<0.044) was adjusted for two interim analyses, and all tests were conducted using two-sided tests; Adjusted Relative Risk = 0.75, 95% CI 2-sided [0.52 to 1.08]

2. Primary Outcome: 30-day Mortality
Time Frame: First 30 days after ED admission
Population: Number of subjects enrolled into each group.
Measure: Number; unit: participants
Arm/Group | 1:1:1 Blood Transfusion Ratio | 1:1:2 Blood Transfusion Ratio
Number analyzed (Participants) | 338 | 342
participants | 75 | 89
Statistical Analysis 1: Comparison: 1:1:1 Blood Transfusion Ratio vs 1:1:2 Blood Transfusion Ratio; Initial sample size of 580 planned to detect clinically meaningful a 12% difference in 30-day mortality (23% vs. 35%),supported by prior data. DSMB increased sample size to 680 according to trial's adaptive design. With 680 patients & given final observed mortality proportions in the 1:1:1 group, PROPPR had 92% power to detect the pre-specified 12% difference at 30 days, if such differences existed; Test type: Superiority or Other; p = 0.26, Mantel Haenszel; [statistical method as in outcome 1, analysis 1]; Adjusted Relative Risk = 0.86, 95% CI 2-sided [0.65 to 1.12]

3. Primary Outcome: Coagulation as Indicated by Number of Participants With Reported Venous Thrombolic Events (VTE)
Description: Blood samples were collected at time of ED admission and over time to determine the incidence of reported venous thrombolic events (VTE).
Time Frame: From time of ED admission, for up to 72 hours
Population: Number of subjects who were randomized to each group
Measure: Number; unit: participants
Groups:
- 1:1:1 Blood Transfusion Ratio: 1:1:1 Blood Transfusion Ratio: Group 1 will be randomized to receive the 1:1:1 ratio.
- 1:1:2 Blood Transfusion Ratio: 1:1:2 Blood Transfusion Ratio: Group 2 will be randomized to receive the 1:1:2 ratio.
Arm/Group | 1:1:1 Blood Transfusion Ratio | 1:1:2 Blood Transfusion Ratio
Number analyzed (Participants) | 338 | 342
participants | 45 | 42

4. Secondary Outcome: Hospital Free Days
Time Frame: first 30 days after ED admission
Population: Number of hospital free days for each group.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | 1:1:1 Blood Transfusion Ratio | 1:1:2 Blood Transfusion Ratio
Number analyzed (Participants) | 338 | 342
days | 1 [0 to 17] | 0 [0 to 16]
Statistical Analysis 1: Comparison: 1:1:1 Blood Transfusion Ratio vs 1:1:2 Blood Transfusion Ratio; Test type: Superiority or Other; p = 0.83, van Elteren's test for medians

5. Secondary Outcome: Time to Hemostasis
Description: Time to hemostasis refers to the time that the subject achieved hemorrhage control (anatomic hemostasis and resuscitation complete)following emergency department (ED) arrival.
Time Frame: ED admission to hospital discharge or 30 days, whichever comes first
Population: Time to anatomic hemostasis
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | 1:1:1 Blood Transfusion Ratio | 1:1:2 Blood Transfusion Ratio
Number analyzed (Participants) | 338 | 342
minutes | 105 [64 to 179] | 100 [56 to 181]
Statistical Analysis 1: Comparison: 1:1:1 Blood Transfusion Ratio vs 1:1:2 Blood Transfusion Ratio; Test type: Superiority or Other; p = 0.44, van Elteren's test for medians

6. Secondary Outcome: Amount of Randomized Blood Products Given to Hemostasis
Time Frame: 24 hours from randomization
Measure: Median (Inter-Quartile Range); unit: units of blood products
Arm/Group | 1:1:1 Blood Transfusion Ratio | 1:1:2 Blood Transfusion Ratio
Number analyzed (Participants) | 338 | 342
units of blood products | 16 [10 to 32] | 15 [5 to 24]

7. Secondary Outcome: Functional Status at Time of Hospital Discharge
Description: The Glasgow Outcome Extended Score (GOSE) is a tool used to measure recovery following brain injury and assists with prediction of long-term rehabilitation. The 8 scoring categories are death, vegetative state, lower severe disability, upper severe disability, lower moderate disability, upper moderate disability, lower good recovery and upper good recovery. A higher GOSE score correlates with better outcome.
Time Frame: Hospital discharge or 30 days, whichever comes first
Population: Glasgow Outcome Extended Score (GOSE) Score on discharged patients who had a head injury (Abbreviated Injury Score (AIS) > 1) ranging from 1 to 8. The AIS is a coding scale to classify the injury severity. A score is created for each body region, type of anatomic structure (i.e. whole area, vessels,organs), and severity(minor to maximum).
Measure: Median (Inter-Quartile Range); unit: units on the GOSE scale
Arm/Group | 1:1:1 Blood Transfusion Ratio | 1:1:2 Blood Transfusion Ratio
Number analyzed (Participants) | 30 | 28
units on the GOSE scale | 4 [3 to 6] | 4.5 [3.5 to 7]
Statistical Analysis 1: Comparison: 1:1:1 Blood Transfusion Ratio vs 1:1:2 Blood Transfusion Ratio; Test type: Superiority or Other; p = 0.11, van Elteren's test for medians

8. Secondary Outcome: Incidence of Primary Surgical Procedure
Time Frame: ED admission to hospital discharge or 30 days, whichever comes first
Population: Incidence of primary surgical procedure
Measure: Number; unit: participants
Arm/Group | 1:1:1 Blood Transfusion Ratio | 1:1:2 Blood Transfusion Ratio
Number analyzed (Participants) | 338 | 342
participants | 290 | 284
Statistical Analysis 1: Comparison: 1:1:1 Blood Transfusion Ratio vs 1:1:2 Blood Transfusion Ratio; Test type: Superiority or Other; Risk Difference (RD) = 2.8, 95% CI 2-sided [-2.8 to 8.3]

9. Secondary Outcome: Incidence of Transfusion Related Serious Adverse Events
Time Frame: ED admission to hospital discharge or 30 days, whichever comes first
Population: Incidence of transfusion related serious adverse events-Reportable to FDA
Measure: Number; unit: participants
Arm/Group | 1:1:1 Blood Transfusion Ratio | 1:1:2 Blood Transfusion Ratio
Number analyzed (Participants) | 338 | 342
participants | 1 | 0
Statistical Analysis 1: Comparison: 1:1:1 Blood Transfusion Ratio vs 1:1:2 Blood Transfusion Ratio; Test type: Superiority or Other; Risk Difference (RD) = 0.3, 95% CI 2-sided [-0.8 to 1.7]

10. Secondary Outcome: Initial Hospital Discharge Status
Time Frame: Hospital discharge or 30 days, whichever comes first
Population: Disposition of subject at time of hospital discharge
Measure: Number; unit: participants
Arm/Group | 1:1:1 Blood Transfusion Ratio | 1:1:2 Blood Transfusion Ratio
Number analyzed (Participants) | 338 | 342
participants
  Home | 118 | 105
  Remained hospitalized at 30 days | 82 | 77
  Other | 59 | 71
  Morgue | 75 | 89
  Unknown | 4 | 0
Statistical Analysis 1: Comparison: 1:1:1 Blood Transfusion Ratio vs 1:1:2 Blood Transfusion Ratio; Test type: Superiority or Other; p = 0.37, generalized logit model regression

11. Secondary Outcome: Ventilator Free Days
Time Frame: first 30 days after ED admission
Population: Number of ventilator free days for each group.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | 1:1:1 Blood Transfusion Ratio | 1:1:2 Blood Transfusion Ratio
Number analyzed (Participants) | 338 | 342
days | 8 [0 to 16] | 7 [0 to 14]
Statistical Analysis 1: Comparison: 1:1:1 Blood Transfusion Ratio vs 1:1:2 Blood Transfusion Ratio; Test type: Superiority or Other; p = 0.14, van Elteren's test for medians

12. Secondary Outcome: ICU Free Days
Time Frame: first 30 days after ED admission
Population: Number of ICU free days for each group.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | 1:1:1 Blood Transfusion Ratio | 1:1:2 Blood Transfusion Ratio
Number analyzed (Participants) | 338 | 342
days | 5 [0 to 11] | 4 [0 to 10]
Statistical Analysis 1: Comparison: 1:1:1 Blood Transfusion Ratio vs 1:1:2 Blood Transfusion Ratio; Test type: Superiority or Other; p = 0.10, van Elteren's test for medians

13. Secondary Outcome: Amount of Blood Products Given From Hemostasis to 24 Hours After ED Admission
Time Frame: 24 hours after ED admission
Population: Unit of measure for outcome measures below is median number of blood product units that given in each group (1:1:1 or 1:1:2) from time initial hemostasis was complete (PROPPR randomized study products stopped) up to 24 hours following ED admission. Number of participants is based on those who survived up to 24 hours, not participants randomized.
Measure: Median (Inter-Quartile Range); unit: units of blood products
Arm/Group | 1:1:1 Blood Transfusion Ratio | 1:1:2 Blood Transfusion Ratio
Number analyzed (Participants) | 316 | 305
units of blood products | 1 [0 to 6] | 2 [0 to 9]

ADVERSE EVENTS:
Time Frame: up to 30 days following ED admission
Arm/Group | 1:1:1 Blood Transfusion Ratio | 1:1:2 Blood Transfusion Ratio
Serious Adverse Events (participants affected / at risk) | 2/338 | 4/342
Other Adverse Events (participants affected / at risk) | 297/338 | 310/342
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1:1:1 Blood Transfusion Ratio (N=338) | 1:1:2 Blood Transfusion Ratio (N=342)
Transfusion-associated circulatory overload (Cardiac disorders) | 1 (1) | 0 (0) — Serious adverse event reportable to FDA
Hypernatremia associated with hypertonic saline use (Metabolism and nutrition disorders) | 1 (1) | 4 (4) — Serious adverse events reportable to FDA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1:1:1 Blood Transfusion Ratio (N=338) | 1:1:2 Blood Transfusion Ratio (N=342)
Systemic inflammatory response syndrome (General disorders) | 231 (265) | 216 (239)
Sepsis (Infections and infestations) | 99 (110) | 91 (102)
Infection (Infections and infestations) | 98 (155) | 106 (146) — Includes urinary tract infection, wound infection, line infection and other. Data is not available for the specific types of infection (i.e. urinary, wound, line).
Acute Kidney Injury (Renal and urinary disorders) | 74 (87) | 85 (93)
Ventilator-associated pneumonia (Infections and infestations) | 62 (70) | 58 (65)
Transfusion-related metabolic complications (Metabolism and nutrition disorders) | 53 (53) | 59 (60) — Hypocalcemia and hyperkalemia only
Acute Lung Injury (Respiratory, thoracic and mediastinal disorders) | 47 (56) | 57 (66)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 46 (55) | 48 (57)
Deep Vein Thrombosis (Vascular disorders) | 25 (28) | 24 (24)
Abdominal Complication (General disorders) | 24 (29) | 22 (23) — Also includes complications related to injury
Cardiac arrest (Cardiac disorders) | 23 (25) | 27 (30)
Multiple Organ Failure (General disorders) | 20 (24) | 15 (18)
Symptomatic pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 13 (13)
Additional bleeding after hemostasis requiring intervention (General disorders) | 13 (13) | 16 (18) — bleeding occurring after hemostasis requiring an interventional radiology or surgical procedure
Asymptomatic pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 11 (11)
Stroke (Nervous system disorders) | 8 (9) | 11 (11)
Abdominal Compartment syndrome (General disorders) | 3 (3) | 3 (3)
Delayed serological transfusion reaction (Immune system disorders) | 2 (2) | 0 (0)
Transfusion-related allergic reaction (General disorders) | 2 (2) | 1 (1)
Febrile nonhemolytic transfusion reaction (Immune system disorders) | 1 (1) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No